CLINICAL TRIAL: NCT05891925
Title: An Audiobook-based Intervention on Community-dwelling Older Adults in Concepción, Chile
Brief Title: An Audiobook-based Intervention on Community-dwelling Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Católica de la Santísima Concepción (Other)
Collaborators: Universidad de Concepcion (Other)
Responsible Party: Principal Investigator, Pedro O. Rossel, Head of the Computer Science Department, Universidad Católica de la Santísima Concepción
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSantísimaConcepción
Record Dates: First submitted 2023-05-12; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Psychological Well-Being; Mental Health
Keywords: older adults; well-being; audiobook; self-care; healthy aging; eHealth
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study will be conducted over 30 older adults who will use an audiobook mobile application for 4 weeks. Participants will be evaluated pre and post intervention through validated questionnaires on digital competences, usability, and perception of well-being.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- older_adults_CRC (Experimental): Over 30 healthy community-dwelling older adults belonging to a Community Rehabilitation Center (CRC) at Concepcion, Chile.
  Interventions: Other: Audiobook App

INTERVENTIONS:
Other: Audiobook App — The intervention will consist of the use of the audiobook application (with poems) for 4 weeks. Here, the application will record the following data autonomously:
  * older adult id,
  * date, hour and time that the older adult listened to each poem,
  * poems listened.
  Initially, two questionnaires will be applied to the older adults: one to measure their digital skills (DIGCOMP), and another to assess their well-being prior to the experience with the audiobook application (Part A).
  After two weeks of application use, a follow-up will be carried out, in order to answer any questions that may arise from the use of the application, and explain again the objectives of the research, if necessary. This follow-up will be initially done by telephone, and in person if required.
  After four weeks, the older adult will be invited to a meeting at the Community Rehabilitation Center at Concepción, Chile, to answer the well-being questionnaire (Part B) and the usability questionnaire (SUS).

SUMMARY:
The goal of this quasiexperimental study is to assess the impact of an audiobook mobile application on the well-being perception of older adults belonging to a Community Rehabilitation Center (CRC) at Concepcion, Chile. The main question is does listening to audio poems using a mobile application improve the perception of well-being of the older adults who go to the CRC at Concepcion? Participants will evaluate the usability of the mobile application designed for this population. The duration of the study will be 4 weeks.

DETAILED DESCRIPTION:
The worldwide population over 60 years of age is increasing. Thus, older adults should maintain interest and participate in social and family activities to help preserve their independence and promote their well-being. Wellbeing is a part of human health in its most general sense which manifests itself in all areas of human activity. Leisure activities such as listening to an audiobook may provide enjoyment and promote relaxation in older people and help improve the well-being of older adults.

A quasiexperimental study to assess the impact of an audiobook mobile application on the well-being perception of older adults and the usability of this application will be conducted during the fourth quarter of 2023. In this study, participants will be compared with themselves at the beginning and at the end of the intervention, that is, a pretest/posttest with a single group.

The first stage corresponds to recruiting community-dwelling older adults, to be done at a community center. With the older adults who agree to participate in the study, the researchers will do the second stage (screening), which consists of determining who can participate in the study by applying the inclusion and exclusion criteria (third stage). Before starting the intervention, participating older adults must accept and sign a written consent (fourth stage). Then, a baseline (fifth stage) will be established by applying standardized and validated tests to the participating older adults, who will then have an induction session to install the application on their smartphones, learn how to use the application and get answers to any questions the participants might have (sixth stage). In the intervention (seventh stage), the participants will use the application for four weeks, with a follow-up at 2 weeks (eighth stage). After these four weeks of application use, the older adults will be evaluated through standardized tests (ninth stage).

The participants will be recruited from the Community Rehabilitation Center (CRC) at Concepcion, Chile. A sample of 60 older adults participated in a similar study to ours. Thus, a non-probabilistic type of sampling will be used for the convenience of the study. In particular, a minimum of 30 participants and a maximum of 60 will be considered to allow obtaining data from the different quintiles and genders within the sample.

Recruitment flyers will be posted on the walls of the CRC to make an open call to all people over 60 being treated at that place. Furthermore, group meetings scheduled by the researchers will be held at the CRC offices to invite older adults to participate in the research. Older adults interested in the study will register by giving their name and telephone number, and will be contacted later by the researchers.

Older adults interested in participating in the study will be contacted by telephone. Then, the study, the objectives of the research and the strategy to be used in the study will be explained to them in a concise and precise way. Furthermore, the researchers will find out if the participants meet the inclusion criteria for the study.

If the older adults refuse to participate, the older adults will be thanked and told there is no harm to them. Otherwise, the older adults will be invited to a meeting at the CRC, on a schedule to be agreed.

During the meeting, the written informed consent will be handed out and explained to them with the support of the consent itself, emphasizing that participation in the study is voluntary, and that the confidentiality of the each participant's personal information will be safeguarded. If the older adult agrees to the consent, it will be signed by them and by the researcher responsible for the research, and the participant will receive a signed copy of the consent.

Then, two questionnaires will be applied to the older adults: one to measure their digital skills (DIGCOMP), and another to assess their well-being prior to the experience with the audiobook application (Part A). This last questionnaire was built by the authors specifically for this application. It consists of two parts, and both the content and face validity were made through by an expert committee, with clinical experience, knowledge in methodological investigation, and disciplinary knowledge in psychology.

Finally, one of the researchers will explain to the older adults how the application works, and answer any questions the participants may have. After the explanation, the audiobook application will be installed on the older adult's smartphone, and the older adult will be provided with a contact telephone number to answer any questions about the operation of the application.

The intervention will consist of the use of the audiobook application for 4 weeks. During this period, the application will record the following data autonomously: older adult id, date, hour and time that the older adult listened to each poem, poems listened. This data will be stored locally and sent to a server for remote storage when the older adult has internet access.

Considering the hypothesis, there is no minimum application frequency of use to be suggested to participants. Thus, older adults should use the audiobook application according to their time availability and their motivation. Furthermore, participants are advised to abstain from any other emotional, social and/or motor training during the intervention period.

After two weeks of application use, a follow-up will be carried out, in order to answer any questions that may arise from the use of the application, and explain again the objectives of the research, if necessary. This follow-up will be initially done by telephone, and in person if required. After four weeks, the older adult will be invited to a meeting at the CRC, on a schedule to be agreed beforehand, to answer the well-being questionnaire (Part B) and the usability questionnaire (SUS). Finally, data analysis will be carried out once the data gathering is finished.

A positive impact on the perception of well-being is expected in older adults who listen to poems through an audiobook mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Person aged 60 and over who belongs to the Community Rehabilitation Center at Concepción, Chile.
* Speak and read Spanish.
* Enabled and capable of approving the informed consent.
* Provide signed informed consent.
* Older adults who have a smartphone where they can run the audiobook mobile application.
* Older adults who are not participating in other emotional, social and/or motor training programs.

Exclusion Criteria:

* Significant psychiatric or medical illness (depressive disorder, delirium, intellectual disability, etc).
* Older adults classified with dependency criteria.
* Illiterate people.
* Presence of a severe sensory deficit, either in visual or hearing difficulties.
* Presence of neurodegenerative diseases (dementia, Alzheimer's disease, Parkinson's disease, multiple sclerosis, etc.).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Well-being perception pre-intervention | Pre intervention (just before the start of the intervention)
  "Well-being questionnaire Part A" is related to well-being perception, and this will measure the well-being of the older adults before the use of the audiobook application. This questionnaire was built by the researchers specifically for this application.
  Part A includes 6 questions that are assessed with a 5-point Likert subjective scale (1 strongly disagree and 5 strongly agree). This questionnaire measures the following types of well-being: Hedonic, Eudaimonic, and Social.
  The score obtained in the questionnaire Part A will be between 6 and 30. This score represents the final well-being obtained for older adults before the use of the application. A higher score mean a better outcome.
Well-being perception post-intervention | Four weeks after the start of the intervention
  "Well-being questionnaire Part B" is related to well-being perception, and this will measure the well-being of the older adults after the use of the audiobook application. This questionnaire was built by the researchers specifically for this application
  Part B includes 12 questions that are assessed with a 5-point Likert subjective scale (1 strongly disagree and 5 strongly agree). This questionnaire measures the following types of well-being: Hedonic, Eudaimonic, and Social.
  The score obtained in the questionnaire Part B will be between 12 and 60. This score represents the final well-being obtained for older adults after the use of the application. A higher score mean a better outcome.
Usability of the Audiobook App | Four weeks after the start of the intervention
  Usability is a software quality attribute that assesses how easy user interfaces are to use.
  To measure the usability of the application, the System Usability Scale (SUS) will be used. It consists of 10 questions that are assessed with a 3-point Likert subjective scale (1 totally disagree and 3 completely agree) and it allows quickly answer. The result is between 0 and 100; the higher the result, the higher the usability level of the application.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Espejo-Videla, Msc, Study Director — Universidad de Concepcion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ki-moon B. Follow-up to the Second World Assembly on Ageing. General Assembly of the United Nations, 2011
- [Background] Wick G, Jansen-Durr P, Berger P, Blasko I, Grubeck-Loebenstein B. Diseases of aging. Vaccine. 2000 Feb 25;18(16):1567-83. doi: 10.1016/s0264-410x(99)00489-2. PMID 10689131
- [Background] Huenchuan-Navarro S. Diferencias Sociales en la Vejez. Aproximaciones Conceptuales y Teóricas. Revista Perspectivas 2003; 12: 13-22.
- [Background] Villafuerte RJ, Alonso AYA, Alonso VY, et al. Elderly well-being and quality of life, a challenge for inter-sectoral action. Medisur. 2017;15(1):85-62.
- [Background] Forsblom, A., Särkämö, T., Laitinen, S., & Tervaniemi, M. The effect of music and audiobook listening on people recovering from stroke: The patient's point of view. Music and Medicine. 2010; 2(4), 229-234.
- [Background] Bauger L, Bongaardt R. Structural developmental psychology and health promotion in the third age. Health Promot Int. 2018 Aug 1;33(4):686-694. doi: 10.1093/heapro/daw104. PMID 28082372
- [Background] Chang Dae Lee, Moon Young Kim, Mi Jung Lee, Jaewon Kang & Erin R. Foster. The relationship between active, balanced participation and well-being in older adults in the United States: A time-use perspective. Journal of Occupational Science. 2023; 30:2, 175-183.
- [Background] Araújo, Lia, Ribeiro, Oscar, & Paúl, Constança. Hedonic and eudaimonic well-being in old age through positive psychology studies: a scoping review. Anales de Psicología. 2017; 33(3), 568-577.
- [Background] Ryan RM, Deci EL. On happiness and human potentials: a review of research on hedonic and eudaimonic well-being. Annu Rev Psychol. 2001;52:141-66. doi: 10.1146/annurev.psych.52.1.141. PMID 11148302
- [Background] Keyes, C. L. M. Social well-being. Social Psychology Quarterly. 1998; 61(2), 121-140.
- [Background] Stav WB, Hallenen T, Lane J, Arbesman M. Systematic review of occupational engagement and health outcomes among community-dwelling older adults. Am J Occup Ther. 2012 May-Jun;66(3):301-10. doi: 10.5014/ajot.2012.003707. PMID 22549595
- [Background] Bauger L, Bongaardt R. The lived experience of well-being in retirement: A phenomenological study. Int J Qual Stud Health Well-being. 2016 Nov 3;11:33110. doi: 10.3402/qhw.v11.33110. eCollection 2016. PMID 27814778
- [Background] Kim J, Lee HY, Christensen MC, Merighi JR. Technology Access and Use, and Their Associations With Social Engagement Among Older Adults: Do Women and Men Differ? J Gerontol B Psychol Sci Soc Sci. 2017 Sep 1;72(5):836-845. doi: 10.1093/geronb/gbw123. PMID 28073816
- [Background] Fang Y, Chau AKC, Wong A, Fung HH, Woo J. Information and communicative technology use enhances psychological well-being of older adults: the roles of age, social connectedness, and frailty status. Aging Ment Health. 2018 Nov;22(11):1516-1524. doi: 10.1080/13607863.2017.1358354. Epub 2017 Aug 4. PMID 28777010
- [Background] Cota T and Ishitani L. Motivation and benefits of digital games for the elderly: a systematic literature review. Revista Brasileira de Computação Aplicada. 2015; 7(1): 2-16.
- [Background] Fletcher, J. & Jensen, R. Mobile health: Barriers to mobile phone use in the aging population. Online Journal of Nursing Informatics (OJNI). 2015; 19 (3): 3-10.
- [Background] Carolyn Pang, Zhiqin Collin Wang, Joanna McGrenere, Rock Leung, Jiamin Dai, and Karyn Moffatt. Technology Adoption and Learning Preferences for Older Adults: Evolving Perceptions, Ongoing Challenges, and Emerging Design Opportunities. In Proceedings of the 2021 CHI Conference on Human Factors in Computing Systems (CHI '21). 2021; Association for Computing Machinery, New York, NY, USA, 18 pages. DOI: https://doi.org/10.1145/3411764.3445702.
- [Background] Wilson J, Heinsch M, Betts D, Booth D, Kay-Lambkin F. Barriers and facilitators to the use of e-health by older adults: a scoping review. BMC Public Health. 2021 Aug 17;21(1):1556. doi: 10.1186/s12889-021-11623-w. PMID 34399716
- [Background] García-Rodríguez A and Gomez-Díaz R. ¿Leer con los oídos?: Audiolibros y literatura infantil y juvenil. Anuario ThinkEPI. 2019; 13: e13c01.
- [Background] Ameri F, Vazifeshenas N, Haghparast A. The Impact of Audio Book on the Elderly Mental Health. Basic Clin Neurosci. 2017 Sep-Oct;8(5):361-370. doi: 10.18869/nirp.bcn.8.5.361. PMID 29167723
- [Background] Deng T,Wu J and ZhangW. Audiobooks in the Post-pandemic Era: How Can Audiobooks Boost the Silver Economy as a Hot Medium. In Proceedings of the 2022 3rd International Conference on Language, Art and Cultural Exchange (ICLACE 2022). Atlantis Press, pp. 768-772.
- [Background] Silva PA, Holden K and Jordan P. Towards a List of Heuristics to Evaluate Smartphone Apps Targeted at Older Adults: A Study with Apps that Aim at Promoting Health and WellBeing. In 48th Hawaii International Conference on System Sciences. IEEE, pp. 3237-3246.
- [Background] Ferrari A. Digital Competence in Practice: An Analysis of Frameworks. Technical Report EUR 25351 EN, Research Centre of the European Commission, 2012.
- [Background] Tsang S, Royse CF, Terkawi AS. Guidelines for developing, translating, and validating a questionnaire in perioperative and pain medicine. Saudi J Anaesth. 2017 May;11(Suppl 1):S80-S89. doi: 10.4103/sja.SJA_203_17. PMID 28616007
- [Background] Brooke J. SUS-A quick and dirty usability scale. Usability Evaluation in Industry 1996; 189(194): 4-7.
- [Background] Poerio, G., Totterdell, P. (2020). The effect of fiction on the well-being of older adults: A longitudinal RCT intervention study using audiobooks. Psychosocial Intervention, 29(1), 29-37.
- [Background] Xue Ning FC, Mai-Sarah Mukari SZ and Ahmad K. The effects of familiar, unfamiliar music and audiobooks exposure on speech parameters of elderly with alzheimer's disease: a within case studies. PEOPLE: International Journal of Social Sciences. 2016; 2(1): 397-414.
- [Derived] Aravena-Canese L, Espejo-Videla V, Rossel PO. How does a poetry audiobook app improve the perception of well-being in older adults? A study protocol. PLoS One. 2024 Oct 31;19(10):e0312463. doi: 10.1371/journal.pone.0312463. eCollection 2024. PMID 39480784
- See also: Instituto Nacional de Estadística (INE) Chile. Demografía y vitales, 2023. — https://www.ine.cl/estadisticas/sociales/demografia-y-vitales
- See also: World Health Organization — https://www.who.int/news-room/facts-in-pictures/detail/ageing